CLINICAL TRIAL: NCT04419623
Title: A Phase 1/2, Double-Blind, Randomized, Placebo-Controlled Study of TL-895 With Standard Available Treatment Versus Standard Available Treatment for the Treatment of COVID-19 in Patients With Cancer
Brief Title: A Study of TL-895 With Standard Available Treatment Versus Standard Available Treatment for the Treatment of COVID-19 in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL-895-202
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: COVID-19; Sars-CoV2; Cancer; Solid Tumor; Carcinoma; Blood Cancer
Keywords: TKI; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — COVID-19; Neoplasms; Carcinoma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Up to 18 subjects will participate in a dose-finding safety lead-in to determine the recommended TL-895 dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Finding - 200mg BID (Experimental): 200mg TL-895 orally BID taken continuously in 7-day cycles for 2 - 4 cycles with SAT for COVID-19 (14 - 28 days of treatment).
  Interventions: Drug: TL-895

INTERVENTIONS:
Drug: TL-895 — TL-895, administered by mouth

SUMMARY:
This study evaluates TL-895, a tyrosine kinase inhibitor (TKI). This is a study comprising a Phase 1 safety assessment. TL-895 open-label will be administered orally at an assigned dose continuously in 7-day cycles for 2 cycles. Up to 3 dose levels will be evaluated.

Only Phase 1 of the study was enrolled and the study did not proceed into Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of active cancer that is not considered cured or disease free.
* Confirmed COVID-19 infection as per World Health Organization (WHO) criteria with suspected pneumonia requiring hospitalization and oxygen saturation < 94% on room air or requires supplemental oxygen.
* Adequate hematological, hepatic and renal function as would be medically expected of a cancer patient population.
* Able to swallow and absorb oral medications.

Exclusion Criteria:

* Current active treatment with medications contraindicated for receipt of investigational product.
* Require chemotherapy or urgent systemic therapy for active cancer that cannot be withheld.
* No remaining available therapies for advanced or metastatic malignancies.
* Participation in another clinical study with therapeutic intent for COVID-19
* Require artificial ventilation at screening.
* Life expectancy less than 6 months.
* Medical conditions that make it unsafe to receive investigational product (for example, heart attack in the last 6 mos, unstable angina, uncontrolled arrhythmia, heart failure class 3/4, QTC interval > 480 msec; known bleeding disorders, stroke or intracranial hemorrhage in the last 6 mos; active HBV, HCV or history of HIV; GI malabsorption syndrome, small bowel resection, poorly controlled IBS; untreated/actively progressing known CNS lesions).
* Receipt of radiation therapy to the lung or mediastinum for treatment of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Recommended dose of TL-895 | After the day 14 of the 6th subject per dose level
  To determine the recommended dose of TL-895 to be based on the observed dose limiting toxicity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgia Cancer Center, Augusta, Georgia
  - The Ohio State Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No